CLINICAL TRIAL: NCT06688201
Title: Minimally Invasive Soft Channel Brain Haemorrhage Evacuation for Acute Basal Ganglia Haemorrhage-- Large Hemorrhage Evacuation (MIRACLE-L)
Acronym: MIRACLE-L
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Linyi People's Hospital (Other); Fudan University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor ,Beijing Institute of Brain Disorders,Captial Medcial University, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIRACLE-L
Record Dates: First submitted 2024-10-17; First posted 2024-11-14 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Other neurosurgical techniques (Other): Those include open craniotomy, small skull window microsurgery, and endoscopic surgery.
  Interventions: Other: Other neurosurgical techniques
- Minimally Invasive Soft Channel Brain Haemorrhage Evacuation (Experimental): Minimally Invasive Soft Channel Brain Haemorrhage Evacuation
  Interventions: Procedure: Minimally Invasive Soft Channel Brain Haemorrhage Evacuation

INTERVENTIONS:
Other: Other neurosurgical techniques — Those include open craniotomy, small skull window microsurgery, and endoscopic surgery. The attending clinician is required to consider which type of craniotomy or other procedure according to the expertise and availability at the hospital.
  Arms: Other neurosurgical techniques
Procedure: Minimally Invasive Soft Channel Brain Haemorrhage Evacuation — This technique is based on the study of hematoma anatomy, cerebral vascular anatomy, and neural fiber structure anatomy in basal ganglia hemorrhage to determine the optimal surgical (catheter insertion) path. By applying stereogeometric principles, it allows for simple yet precise localization. Through surgical steps including puncture, aspiration, liquefaction (intermittent infusion of urokinase or alteplase), and external drainage, the hematoma can be completely removed in stages over a short period. This ensures that hematoma clearance and decompression of the brain occur simultaneously, achieving a minimally invasive intracerebral hemorrhage evacuation technique with a gradual reduction in intracranial pressure.
  Arms: Minimally Invasive Soft Channel Brain Haemorrhage Evacuation

SUMMARY:
To determine if minimally invasive soft channel brain hemorrhage evacuation (scMIS), compared with any other neurosurgical technique that includes open craniotomy, small skull window microsurgery , and endoscopic surgery, is at least as effective ('not inferior') on poor clinical outcome of death or major disability (mRS scores 4-6) at 6 months in basal ganglia intracerebral hemorrhage (ICH) of 30 < volume ≤ 100 ml.

ELIGIBILITY:
* Inclusion Criteria:

  1. Adults (18 - 80 years) ;
  2. The clinical diagnosis is acute intracerebral hemorrhage, confirmed by imaging;
  3. Onset within 48 hours, and surgery can be initiated within 48 hours;
  4. Basal ganglia hemorrhage, with a bleeding volume of 30 < volume ≤ 100 ml;
  5. Reduced level of consciousness (GCS 4-14);
  6. Pre-stroke mRS score≤1 points;
  7. Systolic blood pressure <140 mmHg before randomisation;
  8. Availability of being able to receive either scMIS or other neurosurgical technique;
  9. Informed consent obtain accordingly to local regulations.
* Exclusion Criteria:

  1. Definite evidence the ICH is secondary to a structural abnormality in the brain (eg arteriovenous malformation, intracranial aneurysm, tumour, trauma, cerebral venous thrombosis) or previous thrombolysis or neurointerventional surgery.
  2. A high likelihood that the patient will not adhere to the study treatment and follow-up regimen.
  3. Platelet count < 100,000, INR > 1.4.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2025-01-04 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is death or major disability (mRS scores 0-3) at 6 months. | 6 months after randomization
  Ordinal analysis of modified Rankin Scale [mRS] score: 0 =No symptoms at all.1 =No significant disability despite symptoms, able to carry out all usual duties and activities.2 =Slight disability, unable to carry out all previous activities but able to look after own affairs without assistance.3 =Moderate disability requiring some help, but able to walk without Assistance. 4 =Moderate severe disability, unable to walk without assistance and unable to attend to own bodily needs without assistance.5 =Severe disability, bedridden incontinent, and requiring constant nursing care and attention.6 =Dead.

SECONDARY OUTCOMES:
Discharge at Day 7 (yes vs. no) | 7 days after randomization
  Discharge status will be assessed at Day 7
Total length of intensive care unit stay | During hospitalisation up to 6 months after randomization
  The complete length of time a patient is admitted to the intensive care unit (ICU)
Ordinal analysis of modified Rankin Scale [mRS] scores at 28 days | 28 days after randomization
  Ordinal analysis of modified Rankin Scale [mRS] score: 0 =No symptoms at all.1 =No significant disability despite symptoms, able to carry out all usual duties and activities.2 =Slight disability, unable to carry out all previous activities but able to look after own affairs without assistance.3 =Moderate disability requiring some help, but able to walk without Assistance. 4 =Moderate severe disability, unable to walk without assistance and unable to attend to own bodily needs without assistance.5 =Severe disability, bedridden incontinent, and requiring constant nursing care and attention.6 =Dead.
The following at 6-months: ordinal analysis of modified Rankin Scale [mRS] scores 3-6 | 6-months after randomization
  Proportion of subjects with modified Rankin Scale [mRS] 3-6 at 6 months after randomization.
The following at 6-months: ordinal analysis of modified Rankin Scale [mRS] scores 3-5 | 6-months after randomization
  Modified Rankin Scale [mRS] score at 6 months analysed as an ordinal outcome (categories 3 to 5).
The following at 6-months: ordinal analysis of modified Rankin Scale [mRS] scores 0-6 | 6-months after randomization
  Modified Rankin Scale [mRS] score at 6 months analysed as an ordinal outcome (categories 0 to 6).
The following at 6-months: AMC Linear Disability Score(ALDs) | 6-months after randomization
  The AMC (Academic Medical Center) Linear Disability Score (ALDs) is a calibrated generic item bank designed to measure physical disability levels in patients. The ALDs is a sensitive and generic scale that encompasses a broader range of activities compared to the Rankin assessment. The key distinction between the ALDs and the Rankin assessment is that the ALDs provides a linear disability score based on patient-reported outcomes, while the Rankin score is an ordinal assessment determined by a rater.
The following at 6-months: EuroQoL Group 5-Dimension self-report questionnaire (EQ-5D) | 6-months after randomization
  An EQ-5D score, also referred to as an EQ-5D value index or utility, quantifies a person's health status on a scale from 1 (full health) to 0 (equivalent to being dead). Negative values may be assigned to health states considered worse than death.The score is calculated using a formula that applies specific weights to each level in the various dimensions of the EQ-5D, with these weights derived from a value set that includes index values for all possible EQ-5D states.
Days of hospitalization | During hospitalisation up to 6 months after randomization
  Length of stay in hospital.

OTHER OUTCOMES:
Safety outcomes | Throughout the entire study period up to 6 months after randomization
  Mortality, rebleeding, infections, and other serious adverse events (SAEs) recorded throughout the entire study period.

CONTACTS AND LOCATIONS:
Overall Officials: XunMing Ji, PhD, Principal Investigator — Capital Medical University
Locations (1):
- Linyi People's Hospital, Linyi, Shandong, China

IPD SHARING:
Plan to Share IPD: No